CLINICAL TRIAL: NCT02791685
Title: Smartphone Delivered In-home Cardiopulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amit J. Shah, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00085938; 2025P008772 (Other: Emory IRB)
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Disease; Coronary Artery Disease
Keywords: Cardiac Rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cardiac Rehabilitation - Movn Program (Experimental): Participants with coronary artery disease (CAD) and chronic obstructive pulmonary disease (COPD) who are eligible for cardiac rehabilitation will undergo an in-home program.
  Interventions: Behavioral: MULTIFIT Cardiac Rehabilitation
- Pulmonary Rehabilitation - Movn Program (Experimental): Participants with stable chronic obstructive pulmonary disease (COPD) or hospitalized with an acute exacerbation of COPD will undergo an in-home pulmonary rehabilitation program.
  Interventions: Behavioral: Movn Pulmonary Rehabilitation
- Traditional Cardiac Rehabilitation (Active Comparator): Participants enrolled in a facility's traditional cardiac rehabilitation program will be seen at baseline and during a 12 and 24 week follow-up visit.
  Interventions: Behavioral: Standard of Care Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: MULTIFIT Cardiac Rehabilitation — MULTIFIT is a cardiac rehabilitation program delivered by the Movn smartphone application that will provide risk factor modification, prescribed exercises, education and counseling. The application will track activity using a built-in accelerometer or through connected devices such as a Fitbit for daily physical activity and management. Weight and blood pressure (BP) will be tracked by manual input or through wireless scales and BP monitors. The program will last for 12 weeks.
  Arms: Cardiac Rehabilitation - Movn Program
Behavioral: Movn Pulmonary Rehabilitation — Movn pulmonary rehabilitation is a program delivered by the Movn smartphone application that includes targeted educational content and prescribed exercises with mild resistance training in addition to walking and other cardiovascular exercises. The application will track activity using a built-in accelerometer or through connected devices such as a Fitbit for daily physical activity and management. Weight and blood pressure (BP) will be tracked by manual input or through wireless scales and BP monitors. The program will last for 12 weeks.
  Arms: Pulmonary Rehabilitation - Movn Program
Behavioral: Standard of Care Cardiac Rehabilitation — Standard cardiac rehabilitation involves a facility's standard rehabilitation practices. Participants will be seen at baseline and during a 12 and 24 week follow-up visit.
  Arms: Traditional Cardiac Rehabilitation

SUMMARY:
The goal of this study is to determine if a remote cardiac or pulmonary rehabilitation program delivered via a smartphone application and regular telephone calls will lead to improved delivery of cardiac rehabilitation compared to usual care. This includes increased adherence for eligible veterans, increased program completion, improved patient outcomes as measured by functional capacity, improved patient compliance in monitoring symptoms, improved self-efficacy and knowledge in managing disease and, a decreased rate of hospitalization and re-admissions.

DETAILED DESCRIPTION:
This project aims to determine if a smartphone-delivered cardiac rehabilitation (CR) program could show similar clinical outcomes to in-person programs at a low cost in a large population of patients. Investigators will also assess the feasibility of tailoring a virtual CR program to a small sample of COPD participants who also stand to benefit in the absence of an established pulmonary rehabilitation (PR) program.

This is a non-randomized clinical trial of participants at the Atlanta Veterans Affairs Medical Center with an applicable diagnosis for cardiac or pulmonary rehabilitation versus usual care during the study period. We will evaluate the outcomes related to smartphone-enabled home base cardiopulmonary rehabilitation in those who choose the intervention and those who opt into home-based CR, traditional CR, or those who decline. Data from the past 5 years will also be evaluated to obtain a baseline event rate.

Investigators seek to address the following:

1. Determine whether a home-based cardiac or pulmonary rehabilitation program delivered through smartphones is feasible and improves functional status.
2. Determine if education and lifestyle counseling lead to increased adherence with prescribed follow-up, pharmacotherapy, quality of life, self-efficacy and lifestyle changes.
3. Determine if a home-based cardiac or pulmonary rehabilitation program reduces health system utilization, including ED visits and readmission rates.

ELIGIBILITY:
Inclusion Criteria:

Meet eligibility for cardiac rehabilitation program as defined by Centers for Medicare & Medicaid Services (CMS); they may also have stable CAD and be referred for cardiac rehab by their provider.

1. Following acute myocardial infarction (within the preceding 12 months)
2. Coronary artery bypass grafting (CABG)
3. Current stable angina pectoris
4. Heart valve repair or replacement
5. Percutaneous transluminal coronary angioplasty (PTCA) or coronary stenting
6. Heart or heart-lung transplant
7. Other diagnosis by specific physician referral

Exclusion Criteria:

* Unstable angina
* Resting systolic blood pressure >200 mm Hg or resting diastolic blood pressure >110 mm Hg
* Significant drop (>=20 mm Hg) in resting systolic blood pressure from the patient's average level that cannot be explained by medications
* Moderate to severe aortic stenosis
* Acute systemic illness or fever
* Uncontrolled atrial or ventricular arrhythmias
* Symptomatic congestive heart failure (stage C)
* Third-degree heart block without pacemaker
* Active pericarditis or myocarditis
* Recent venous thromboembolism (VTE, as determined by physician)
* Current Thrombophlebitis
* Uncontrolled diabetes (A1c > 7.0 or as determined by physician)
* Orthopedic problems that would prohibit exercise
* Other by specific physician instruction
* Peripheral vascular disease (PVD; symptomatic or that would prohibit exercise)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2016-05; Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Change in Functional Capacity assessed by the Six Minute Walk Test (6MWT) | Week 12, Week 24
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.

SECONDARY OUTCOMES:
Change in Measure of Exercise Intensity (MET) | Baseline, Week 12
  An exercise test will be used to collect MET.
Change in Weight | Baseline, Week 12
  Weight will be measured in kilograms.
Change in Body Mass Index (BMI) | Baseline, Week 12
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness.
Change in Blood Pressure | Baseline, Week 12
  Blood pressure is measured using a blood pressure cuff to the upper extremity. The top number, which is also the higher of the two numbers, measures the pressure in the arteries when the heart beats (systolic).The bottom number, which is also the lower of the two numbers, measures the pressure in the arteries between heartbeats (diastolic). Readings are measured as follows:
  Normal = systolic less than 120 and diastolic less than 80 Prehypertension = systolic 120 - 139 or diastolic 80 - 89 High Blood Pressure (Hypertension) Stage 1 = systolic 140 - 159 or diastolic 90 - 99 High Blood Pressure(Hypertension) Stage 2 = systolic 160 or higher or diastolic 100 or higher Hypertensive Crisis (Emergency care needed) systolic = higher than 180 or diastolic higher than 110
Change in A1c Level | Baseline, Week 12
  The A1C test is a blood test that provides information about a person's average levels of blood glucose, also called blood sugar, over the past 3 months.
  Levels are measured as follows:
  Normal = below 5.7 percent Diabetes = 6.5 percent or above Prediabetes = 5.7 to 6.4 percent
Change in Low-density Lipoprotein (LDL) Level | Baseline, Week 12
  LDL cholesterol is considered "bad" cholesterol because it contributes to plaque, a thick, hard deposit that can clog arteries and make them less flexible.
  Levels are measured as follows:
  < 100 mg/ dL = Optimal 100-129 mg/dL = Near optimal/above optimal 130-159 mg/dL = Borderline high 160-189 mg/dL = High >190 mg/dL = Very high
Change in Duke Activity Status Index (DASI) Score | Baseline, Week 12
  The Duke Activity Status Index (DASI) is a 12-item questionnaire that utilizes self-reported physical work capacity to estimate peak metabolic equivalents. The DASI is scored by adding all activities performed together. A higher score indicates the ability to perform more physical activities.
Change in Patient Health Questionnaire (PHQ-9) Score | Baseline, Week 12
  The PHQ-9 is an instrument for screening, diagnosing, monitoring, and measuring the severity of depression.
  Score ranges from 5-9 indicate minimal depressive symptoms. Scores 10-14 may indicate minor depression, dysthymia, and mild major depression. Scores 15-19 indicate moderately severe, major depression. Scores greater than or equal to 20 indicate severe major depression.

CONTACTS AND LOCATIONS:
Overall Officials: Amit J Shah, MD, Principal Investigator — Emory University
Locations (1):
- Atlanta VA Medical Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harzand A, Alrohaibani A, Idris MY, Spence H, Parrish CG, Rout PK, Nazar R, Davis-Watts ML, Wright PP, Vakili AA, Abdelhamid S, Vathsangam H, Adesanya A, Park LG, Whooley MA, Wenger NK, Zafari AM, Shah AJ. Effects of a patient-centered digital health intervention in patients referred to cardiac rehabilitation: the Smart HEART clinical trial. BMC Cardiovasc Disord. 2023 Sep 12;23(1):453. doi: 10.1186/s12872-023-03471-w. PMID 37700245
- [Derived] Harzand A, Witbrodt B, Davis-Watts ML, Alrohaibani A, Goese D, Wenger NK, Shah AJ, Zafari AM. Feasibility of a Smartphone-enabled Cardiac Rehabilitation Program in Male Veterans With Previous Clinical Evidence of Coronary Heart Disease. Am J Cardiol. 2018 Nov 1;122(9):1471-1476. doi: 10.1016/j.amjcard.2018.07.028. Epub 2018 Aug 4. PMID 30217377

DOCUMENTS (1):
  • Informed Consent Form (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT02791685/ICF_001.pdf